CLINICAL TRIAL: NCT04904042
Title: Phase I/II Study of Efficiency and Single-arm Safety on the Use of Neutral Argon Plasma in Cyto-reduction of Miliary Implants in the Peritoneal Surface.
Brief Title: Study of Safety and Efficiency of the Use of Neutral Argon Plasma in Cyto-reduction of Miliary Implants in the Peritoneal Surface.
Acronym: Plasmajet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FCO-PLASM-2020-01
Record Dates: First submitted 2021-05-18; First posted 2021-05-27 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Peritoneal carcinomatosis; Cancer; Neutral argon plasma
MeSH Terms: conditions — Peritoneal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of plasma of neutral argon (Experimental): Use of plasma of neutral argon in the eradication of tumor implants at the mesentery level, with different doses (established according to the percentage of energy used) and distances of application and time. It will also be compared in-vivo with control therapy of Monopolar electrofulguration at a power of 100 in cut mode with ball-tip terminal.
  Interventions: Device: Use of plasma of neutral argon

INTERVENTIONS:
Device: Use of plasma of neutral argon — Evaluation of the mesentery or peritoneum area infiltrated by miliary implants that is going to be treated. Determination of the PCI. Collection of several samples of the mesenteric peritoneum or parietal peritoneum with tumor involvement (implants between 1-2.5mm of diameter).
  It will established a matrix which will be divided into 12 quadrants where the tissue with implants will be placed and it will be treated according to specific power (80-100%), and for an action time of 2-4 seconds or until macroscopic tumor destruction. For each power, application of Plasmajet at 1, 2 and 3 cm from the target tumor tissue.
  The in-vivo effect will be evaluated with the use of ball-tip in terms of damage to the serosa or vascularization of the mesentery.

SUMMARY:
Neutral argon plasma vaporization shows little damage to normal tissue and allows a complete removal of tumor tissue, that is, without leaving any cell debris viable tumor.

Our primary objective is to evaluate the effectiveness and safety of neutral argon plasma on peritoneal implants with different dosimetry in vivo and ex vivo.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with peritoneal carcinomatosis (an attempt will be made to cover all histological types of carcinomatosis in similar distribution as 2 patients with carcinomatosis of colonic origin, 2 patients with carcinomatosis of ovarian origin, 2 patients with peritoneal pseudomyxoma, 2 patients with peritoneal mesothelioma and 2 patients with carcinomatosis of gastric origin) with PCI greater than 0 in regions 10-13, and that have been selected as candidates for cytoreductive surgery + HIPEC or for laparoscopy-laparotomy explorer (selection criteria established according to clinical practice usual), and that present peritoneal miliary dissemination consistent with the characteristics of this study for the tissue under examination (implants smaller than 0.25 cm, CC1).
* Signature of specific informed consent for participation in this study and to obtain biological samples.

Exclusion Criteria:

* Patients not suitable for CRS and HIPEC, according to the clinical criteria of the Surgery Unit Oncology and multidisciplinary committee.
* Refusal of the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Pathological evaluation | Through study completion, an average of 1 year.
  Pathological evaluation, in the Pathological Anatomy service of the University Hospital Reina Sofía, of both samples of peritoneum and evaluation of the presence of cells tumors and degree of tissue destruction, after performing the procedure according to the indications of the "Interventions" section.
  The specimens will be fixed in formaldehyde for about 48 hours and cut and fixed in paraffin. They will be stained with hematoxylin and eosin according to protocol, after being cut in the area of greatest macroscopic lesion produced by the device. It will be used microscopy and optical micrometer to measure the depth of vaporization of the tissue, as well as damage to adjacent healthy tissue.
  Depth is measured from a line parallel to the surrounding tissue to the point deeper tissue evaporation. As all quadrants will include tumor implants, they will also have flat tissue without tumor and it will be which the depth is measured from.

SECONDARY OUTCOMES:
Evaluation of mesentery vascular damage and damage to the intestinal serosa. | During the surgery and through study completion, an average of 1 year.
  Evaluation of mesentery vascular damage and damage to the intestinal serosa. It will be evaluated in-vivo and it will be analyzed by a third party on video.
Morbidity associated with treatment. | 30 days after the intervention
  Evaluation of morbidity associated with treatment. Using CTCAE scale v4.0 30 days after the intervention. We will pay special attention to events associated with hemoperitoneum, intestinal fistulas or intestinal perforations.
Mortality associated with treatment. | 30 days after the intervention
  Evaluation of mortality associated with treatment. Using CTCAE scale v4.0 30 days after the intervention. We will pay special attention to events associated with hemoperitoneum, intestinal fistulas or intestinal perforations.
Global morbidity. | Within the 30 days post-intervention
  Evaluation of global morbidity using CTCAE v 4.0 scale.
Global mortality. | Within the 30 days post-intervention
  Evaluation of global mortality using CTCAE v 4.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Arjona-Sanchez, PhD, Principal Investigator — University Hospital Reina Sofia
Locations (1):
- University Hospital Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the conclusion of the study and the results were published
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the publication of the results
Access Criteria: upon request to the principal investigator

REFERENCES:
- [Derived] Pontes-Garcia A, Martinez-Lopez A, Rodriguez-Ortiz L, Valenzuela-Molina F, Rufian-Andujar B, Sanchez-Hidalgo JM, Casado-Adam A, Gordon-Suarez A, Rufian-Pena S, Vazquez-Borrego MC, Romero-Ruiz A, Arjona-Sanchez A. Establishment of a desirable dose using neutral argon plasma to eradicate miliary peritoneal implants: A phase I/II controlled trial. Eur J Surg Oncol. 2023 Sep;49(9):106978. doi: 10.1016/j.ejso.2023.07.004. Epub 2023 Jul 11. PMID 37460370